CLINICAL TRIAL: NCT02883478
Title: A Randomized Study of Clinical and Structural Outcome of Corneal Collagen Crosslinking (CXL) With Conventional Versus Accelerated Ultraviolet-A Irradiation Using Riboflavin With Hydroxypropyl Methylcellulose (HPMC).
Brief Title: Clinical and Structural Outcome of Conventional Versus Accelerated Corneal Collagen Cross-linking (CXL).
Acronym: CXL
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Anne Marie Hagem, MD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010/626 C S-08344c
Record Dates: First submitted 2016-05-30; First posted 2016-08-30 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Keratoconus; Corneal Ectasia
MeSH Terms: conditions — Keratoconus | interventions — Radiotherapy; Radiation; Riboflavin; Hypromellose Derivatives

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment group A (Active Comparator): Corneal collagen cross-linking using riboflavin with hydroxypropyl methylcellulose solution and ultraviolet-A (UVA) irradiation at 3 milliwatt/cm² (mW/cm²) for 30 minutes.
  Device: UV-X 1000 irradiator (3 mW/cm²) Drug: riboflavin with hydroxypropyl methylcellulose
  Interventions: Device: UV-X 1000 (3 mW/cm²); Drug: riboflavin with hydroxypropyl methylcellulose
- Treatment group B (Active Comparator): Corneal collagen cross-linking using riboflavin with hydroxypropyl methylcellulose solution and ultraviolet-A (UVA) irradiation at 9 mW/cm² for 10 minutes.
  Device: UV-X 2000 irradiator (9 mW/cm²) Drug: riboflavin with hydroxypropyl methylcellulose
  Interventions: Procedure: UV-X 2000 (9 mW/cm²); Drug: riboflavin with hydroxypropyl methylcellulose

INTERVENTIONS:
Device: UV-X 1000 (3 mW/cm²) — Ultraviolet-A (UVA) irradiation for 30 minutes at 3 milliwatt/cm² (mW/cm²).
  Other Names: conventional ultraviolet-A(UVA) irradiation
  Arms: Treatment group A
Procedure: UV-X 2000 (9 mW/cm²) — Ultraviolet-A (UVA) irradiation for 10 minutes at 9 mW/cm².
  Other Names: accelerated ultraviolet-A(UVA) irradiation
  Arms: Treatment group B
Drug: riboflavin with hydroxypropyl methylcellulose — Drops of riboflavin with hydroxypropyl methylcellulose will be applied in the eye for 20 minutes before ultraviolet-A(UVA) irradiation and every 2 minutes during UVA irradiation
  Other Names: riboflavin with HPMC

SUMMARY:
Compare different corneal parameters and visual outcome of corneal collagen cross-linking (CXL) with conventional versus accelerated ultraviolet-A irradiation using riboflavin with hydroxypropyl methylcellulose.

DETAILED DESCRIPTION:
40 patients with signs of progressive keratoconus are randomized to either corneal collagen cross-linking (CXL) with conventional ultraviolet-A (UVA) irradiation at 3 milliwatt/cm² (mW/ cm²) or accelerated ultraviolet-A (UVA) irradiation at 9 mW/ cm². In both groups riboflavin with hydroxypropyl methylcellulose was used. The objectives of this study are to evaluate and compare different corneal parameters (maximum corneal curvature, depth of collagen cross-linking, endothelial cell density) and clinical outcomes of uncorrected visual acuity (UCVA) and best spectacle corrected visual acuity (BSCVA)) after CXL with conventional and accelerated UVA irradiation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with increase of minimum of 1,0 diopter in maximum keratometry.
* Patients with increase in corneal astigmatism of minimum 1,0 diopter.
* Patients with in spherical equivalent of min 0,5 diopter.
* Patients living in Eastern Norway.

Exclusion Criteria:

* Minimum pachymetric corneal thickness (Pentacam)<360 µm.
* Central corneal scar.
* Chemical burn, serious corneal infections and ocular surface diseases.
* Pregnancy.
* Lactation.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Compare change in maximum corneal curvature, visual acuity, endothelial cell density and depth of cross-linking in CXL with conventional versus accelerated UVA irradiation. | 2 years
  Compare change in maximum corneal curvature (Kmax; diopter), uncorrected visual acuity (UCVA, logMAR), best spectacle corrected visual acuity (BSCVA, logMAR) from baseline and depth in micrometer(µm) of corneal collagen cross-linking on anterior segment optical coherence tomography and confocal microscopy in corneal collagen cross-linking with conventional at 3 milliwatt/cm² (mW/cm²) versus accelerated (9 mW/cm²) ultraviolet-A irradiation using riboflavin with hydroxypropyl methylcellulose.

SECONDARY OUTCOMES:
Compare depth of corneal collagen cross-linking on anterior segment optical coherence tomography and confocal microscopy with change in endothelial cell density in CXL with conventional versus accelerated ultraviolet-A irradiation. | 2 years
  Compare depth (µm) of corneal collagen cross-linking on anterior segment optical coherence tomography and confocal microscopy with change in endothelial cell density (ECD; cells/mm²) from baseline in CXL with conventional (3 mW/cm²) versus accelerated (9 mW/cm²) ultraviolet-A irradiation using riboflavin with hydroxypropyl methylcellulose..
Compare depth of corneal collagen cross-linking on anterior segment optical coherence tomography and confocal microscopy with change in maximal corneal curvature (Kmax) and visual acuity in CXL with conventional versus accelerated UVA irradiation. | 2 years
  Compare depth (µm) of corneal collagen crosslinking on anterior segment optical coherence tomography and confocal microscopy with change in maximal corneal curvature (Kmax; diopter), uncorrected visual acuity (UCVA, logMAR) and best spectacle corrected visual acuity (BSCVA, logMAR) from baseline in CXL with conventional (3 mW/cm²) versus accelerated (9 mW/cm²) ultraviolet-A irradiation using riboflavin with hydroxypropyl methylcellulose.

IPD SHARING:
Plan to Share IPD: No